CLINICAL TRIAL: NCT00360087
Title: Long-Term, Open-Label, Multicenter, Extension Study of Bosentan in Patients With Pulmonary Hypertension Associated With Sickle Cell Disease Completing a Double-Blind ASSET Study (AC-052-368 or AC 052-369)
Brief Title: A Study of Patients Having Pulmonary Hypertension Associated With Sickle Cell Disease and Completing an ASSET Study
Acronym: ASSET-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Actelion (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor, Actelion
Purpose: Treatment
Other Study IDs: AC-052-371
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Hypertension; Sickle Cell Anemia
Keywords: Treatment Study; Sickle Cell Anemia; 6-Minute Walk; Right Heart Catheterization; Tracleer; Sickle Cell; SCD
MeSH Terms: conditions — Hypertension, Pulmonary; Anemia, Sickle Cell | interventions — Bosentan

INTERVENTIONS:
Drug: Bosentan

SUMMARY:
This study will assess the safety and efficacy of bosentan therapy (in a study known as ASSET) for patients who have high blood pressure in the lungs associated with sickle cell disease. That form of hypertension places people at risk for complications, including shortness of breath, pain, pneumonia, and death. Previous studies have shown that bosentan can be helpful in reducing pulmonary hypertension.

Patients ages 16 and older who have completed the 16-week treatment in the ASSET 1 or ASSET 2 study and who are not pregnant or breastfeeding may be eligible for this study. The research will be conducted in about 25 hospitals in the United States and Europe. Up to 30 participants will be enrolled. The screening visit will involve a physical examination, blood sample of about 3 teaspoons for laboratory tests, and a pregnancy test. Patients' doctors will give them bosentan tablets (62.5 mg each), to take one in the morning and one in the evening. After 1 month, patients will be told whether the dose should be increased to 125 mg tablets to take twice a day. Two weeks after the increase in dose, a blood test will be done to analyze the drug's effects on the liver. After the start of treatment, patients will return for visits every 6 months, when there will be a 6-minute walking test to measure exercise capacity and evaluate shortness of breath. There will be follow-up for patients up to the end of the study and for 28 days after the last dose of bosentan is taken, to collect information about side effects.

Some patients on bosentan have had changes in liver function and red blood cell count. Side effects commonly reported are headache, flushed appearance, inflammation of the throat and nasal passages, and gastrointestinal symptoms. If patients have sudden worsening in breathing in the first few weeks after taking bosentan, they should immediately tell their doctors, because it may be necessary to change the treatment.

DETAILED DESCRIPTION:
The object of this study is to assess long-term safety, tolerability and efficacy of bosentan in patients with pulmonary hypertension (PH) associated with sickle cell disease (SCD). The study population will include male and female patients with sickle cell disease (SS,S-beta-Thalassemia) who have previously completed the 16-week treatment period of the double-blind study of bosentan (ASSET 1 or ASSET 2). Patients who meet all the inclusion criteria and none of the exclusion criteria will be started on 62.5 mg bid for 4 weeks and then start the maintenance dose of 125 mg bid (or stay on 62.5 mg if their weight is less than 40kg/90lbs). Patients will be divided into two groups. Group A will consist of patients who begin this study within 4 weeks of completing ASSET 1 or ASSET2. Group B will consist of patients who begin this study longer than 4 weeks after completing ASSET I or ASSET 2. Patients will remain on drug until the FDA approves the drug for use in patients with pulmonary hypertension or until the sponsor decides to stop the study.

ELIGIBILITY:
* INCLUSION CRITERIA
* Completion of the 16-week treatment period in the double-blind ASSET study
* Women of childbearing potential must have a negative result on their serum pregnancy test and use reliable methods of contraception during study treatment and for 3 months after study treatment termination.

Reliable methods of contraception are:

1. Barrier type devices (e.g., female condom, diaphragm, contraceptive sponge) only in combination with a spermicide.
2. Intra-uterine devices.
3. Oral, injectable, transdermal or implantable contraceptives only in combination with a barrier method.

Hormone-based contraceptives alone, regardless of the route of administration, are not considered to be reliable methods of contraception.

Abstention, rhythm method, and contraception by the partner alone are not acceptable methods of contraception.

Women not of childbearing potential are defined as prepubescent, postmenopausal (i.e., amenorrhea for at least 1 year), or surgically or naturally sterile.

Signed written informed consent is obtained from the patient or patient's parent/ legal representative prior to initiation of any study-related procedure.

EXCLUSION CRITERIA

All patients (Groups A and B):

1. Any major protocol violation in the preceding double-blind ASSET study*.
2. Hemoglobin concentration less than 6.0 g/dL.
3. Pregnancy or breast-feeding.

   * Protocol violations will be reviewed by the monitor during site visits and discussed with the study staff on an ongoing basis and at the patient's completion of the double-blind study.

   Group B only:
4. Acute liver disease.
5. Newly diagnosed cirrhosis or portal hypertension.
6. ALT greater than or equal to 3 times ULN and/or albumin greater than 20% below LLN.
7. Newly diagnosed psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with study requirements.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236
Dates: Start 2006-03; Primary Completion 2007-08 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to all assessed time points in 6MWT, in Borg dyspnea index, and in modified NYHA functional class.

REFERENCES:
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486
- [Background] Castro O, Hoque M, Brown BD. Pulmonary hypertension in sickle cell disease: cardiac catheterization results and survival. Blood. 2003 Feb 15;101(4):1257-61. doi: 10.1182/blood-2002-03-0948. Epub 2002 Oct 3. PMID 12393669
- [Background] Minter KR, Gladwin MT. Pulmonary complications of sickle cell anemia. A need for increased recognition, treatment, and research. Am J Respir Crit Care Med. 2001 Dec 1;164(11):2016-9. doi: 10.1164/ajrccm.164.11.2104101. No abstract available. PMID 11739128
- [Derived] Barst RJ, Mubarak KK, Machado RF, Ataga KI, Benza RL, Castro O, Naeije R, Sood N, Swerdlow PS, Hildesheim M, Gladwin MT; ASSET study group*. Exercise capacity and haemodynamics in patients with sickle cell disease with pulmonary hypertension treated with bosentan: results of the ASSET studies. Br J Haematol. 2010 May;149(3):426-35. doi: 10.1111/j.1365-2141.2010.08097.x. Epub 2010 Feb 17. PMID 20175775
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2006-H-0220.html